CLINICAL TRIAL: NCT02911337
Title: Weight Loss as Therapy for Heart Failure With Preserved Ejection Fraction
Acronym: WTLSSCHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WTLSSCHF
Record Dates: First submitted 2015-07-23; First posted 2016-09-22 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure, Diastolic; Weight Loss
MeSH Terms: conditions — Heart Failure, Diastolic; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle modification (Experimental): Lifestyle modification
  Interventions: Dietary Supplement: lifestyle modification

INTERVENTIONS:
Dietary Supplement: lifestyle modification — Subjects will be given meal replacements (shakes and bars) to be consumed twice per day for 8 weeks, and then once per day for an additional 3 weeks, and then transitioned to a structured diet.

SUMMARY:
The purpose of this study is to examine the efficacy of an intensive, supervised, lifestyle modification program on symptoms and signs of heart failure as well as laboratory and echocardiographic measures of cardiac structure and function. This will be a 6 month trial in 50 patients with a clinical diagnosis of heart failure with preserved ejection fraction (HFpEF). Patients will be enrolled in the Medical University of South Carolina weight management 15 week lifestyle change program which will involve weekly visits that rotate among the clinical specialities (dietary, exercise and behavioral) and scheduled visits with the research Registered Nurse. Each patients baseline data will be used as the control and compared with the same measurements at the 6 month end point.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30
* Able to perform 6 minute hall walk test
* Left Ventricular ejection fraction >45%
* Diagnosis of heart failure with preserved ejection fraction (HFpEF) ; confirmation of HFpEF based on 1 major or 3 minor criteria listed below.

Major:

1. Elevated BNP >200
2. cardiogenic pulmonary edema
3. Pulmonary capillary wedge pressure at rest >15 mmhg or with exercise >25 mmhg using invasive right heart pressure measurement

Minor:

1. Left atrial enlargement (volume >68 ml)
2. increased left ventricular wall thickness (>1.1cm) by echocardiography
3. E/e' >15
4. intermediate level of BNP, 60-199

Exclusion Criteria:

* uncontrolled blood pressure
* severe chronic obstructive pulmonary disease (oxygen or steroid dependent)
* recurrent major depression. presence or history of suicide behavior, and current substantial depressive symptoms. Antidepressant drugs are allowed if the dose has been stable for 3 months
* other major psychiatric illness (schizophrenia, bipolar, dementia)
* significant hepatic dysfunction
* untreated hypothyroidism or hyperthyroidism
* history of drug or alcohol abuse or dependency within the past 12 months
* acute coronary syndrome without revascularization in the past 12 months
* acute coronary syndrome with revascularization in the past 6 months
* Cerebrovascular accident or transient ischemic attack in the past 6 months
* cancer or terminal illness with life expectancy < 3 years
* history of medical noncompliance
* significant anemia (hgb <9)
* life threatening or uncontrolled arrhythmia
* hemodynamically relevant valvular heart disease
* infiltrative heart disease including cardiac amyloidosis, sarcoidosis, Fabry's disease
* genetic hypertrophic cardiomyopathy
* significant pericardial disease
* clinically relevant neuromuscular disease
* pregnant or may become pregnant in the next 6 months
* prior major organ transplant or intent to transplant ( on the transplant list)
* pacemaker dependant
* clinically significant congenital heart disease that may be cause of symptoms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Change in 6 minute hall walk test from baseline | 6 months
  Exercise capacity
Change in symptoms measured with the Minnesota Living With Heart Failure(MLWHF) scores | 6 months
  Quality of life assessment specific for congestive heart failure

SECONDARY OUTCOMES:
Left Ventricular mass | 6 months
  Changes in left ventricular mass will be measured by transthoracic echocardiography
Brain Natriuretic Peptide | 6 months
  Brain natriuretic peptide will be measured in serum using standard commercial assay

OTHER OUTCOMES:
Left Atrial Volume | 6 months
  Left atrial volume will be measured by transthoracic echocardiography
Early mitral inflow velocity/mitral annular velocity (E/e') | 6 months
  E/e' will be measured by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- MUSC Gazes Research Institue, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Hajj EC, El Hajj MC, Sykes B, Lamicq M, Zile MR, Malcolm R, O'Neil PM, Litwin SE. Pragmatic Weight Management Program for Patients With Obesity and Heart Failure With Preserved Ejection Fraction. J Am Heart Assoc. 2021 Nov 2;10(21):e022930. doi: 10.1161/JAHA.121.022930. Epub 2021 Oct 29. PMID 34713711